CLINICAL TRIAL: NCT00633399
Title: A Three-phase Study Designed to Test the Efficacy, Tolerability and Safety of the Combination of Ziprasidone With Selective Serotonin Reuptake Inhibitors (SSRI) for Patients With Major Depressive Disorder (MDD) That do Not Sufficiently Respond to Treatment With SSRIs.
Brief Title: Ziprasidone Augmentation of SSRIs for Patients With Major Depressive Disorder (MDD) That do Not Sufficiently Respond to Treatment With SSRIs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, George I. Papakostas, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-P-002361
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-06

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Major Depression; Depression; Geodon; Ziprasidone; SSRI Augmentation; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder, Treatment-Resistant | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients in group 1 will receive Ziprasidone for the full 8 weeks of Phase 2. If they are in remission following phase two, and decide to enter phase three, they will continue on Ziprasidone for 12 months.
  Interventions: Drug: Ziprasidone
- 2 (Placebo Comparator): Patients in group 2 will receive Placebo for the full 8 weeks of Phase 2. If they are in remission following phase two, and decide to enter phase three, they will continue on Placebo for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ziprasidone — 20mg-80mg a day. Dose increases of 20mg per day may occur at three study visits as directed by clinician. Maximum; 80mg per day per patient.
  Other Names: Geodon
  Arms: 1
Drug: Placebo — 0mg Placebo per day (1-4 tablets per day). "Dose increases" and "dose decreases" may occur, but patient will remain at 0mg placebo.
  Arms: 2

SUMMARY:
The purpose of this study is to see if adding the study drug, ziprasidone, to an antidepressant medication helps improve symptoms of Major Depressive Disorder (MDD). We are studying the drug's effectiveness in treating depression, as well as its safety when it is added to another drug.

Hypothesis A: There will be a difference in the percentage of responders in the two treatment conditions during phase 2; response rates will be higher for the ziprasidone group.

DETAILED DESCRIPTION:
The proposed study involves three phases. The first phase is an 8-week, open-label trial of an SSRI for MDD. Patients who do not experience sufficient symptom improvement following this open-label trial will be enrolled in a 6-week, double-blind, placebo controlled trial of ziprasidone augmentation (second phase). Ziprasidone and placebo-remitters will then enter a 12-month, double-blind extension phase (third phase). We estimate that approximately 400 patients will enter phase 1 of the study so that a minimum of 180 subjects will enter double-blind treatment (phase 2) over 5 years. Each treatment arm during phase 2 will have 90 subjects.

Hypothesis B1: During phase 2, there will be a difference between the two groups in the percentage of responders (50% or greater reduction in symptom severity) with regards to anxious symptoms of MDD as measured by the 14-item Hamilton Anxiety Rating Scale (HAM-A); response rates will be higher for the ziprasidone group.

Hypothesis B2: During phase 2, there will be a difference between the two groups in the percentage of responders (50% or greater reduction in symptom severity) with regards to painful symptoms of MDD, as measured by the overall visual analogue pain (VAS-pain) scale scores; response rates will be higher for the ziprasidone group.

Hypothesis C: The time to relapse during phase 3 will be shorter among adjunctive placebo- than ziprasidone-remitters.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Men or women, 18-65 years of age.
* MDD, current, according to DSM-IV criteria and as diagnosed by the SCID- I/P during the screen and baseline visit of phase 1.
* A HAM-D-17 score > 14 during the screen and baseline visit of phase 1.

Exclusion Criteria:

* Pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (oral contraceptive or implant, condom, diaphragm, spermicide, intrauterine
* Device, tubal ligation, or partner with vasectomy).
* Serious suicide or homicide risk, as assessed by evaluating clinician.
* Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease or uncontrolled seizure disorder.
* History of multiple adverse drug reactions or allergy to the study drug.
* The following DSM-IV diagnoses: substance use disorders active within the last six months, any bipolar disorder (current or past), any psychotic disorder (current or past).
* Patients requiring excluded medications (see appendix 1 for details).
* Psychotic features in the current episode or a history of psychotic features.
* Prior course of ziprasidone, or intolerance to ziprasidone at any dose.
* Any investigational psychotropic drug within the last 3 months.
* Have failed more than 3 adequate antidepressant trials during the current MDE. Some examples of adequate dosage of an antidepressant trial include either > 150 mg of imipramine (or its tricyclic equivalent), > 60 mg of phenelzine (or its monoamine oxidase inhibitor equivalent), > 20 mg of fluoxetine (or its SSRI-equivalent), > 150mg of bupropion, > 300mg of trazodone (or nefazodone), >75 mg of venlafaxine, >60mg of duloxetine, or > 15mg of mirtazapine. A trial of adequate duration was defined as one during which the patient was on any given antidepressant at an adequate dose for a minimum of 6 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2008-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George I Papakostas, M.D., Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Massachusetts General Hospital- Depression Clinical and Research Program, Boston, Massachusetts

REFERENCES:
- [Derived] Mischoulon D, Shelton RC, Baer L, Bobo WV, Curren L, Fava M, Papakostas GI. Ziprasidone Augmentation of Escitalopram for Major Depressive Disorder: Cardiac, Endocrine, Metabolic, and Motoric Effects in a Randomized, Double-Blind, Placebo-Controlled Study. J Clin Psychiatry. 2017 Apr;78(4):449-455. doi: 10.4088/JCP.15m10426. PMID 27835715
- [Derived] Ionescu DF, Shelton RC, Baer L, Meade KH, Swee MB, Fava M, Papakostas GI. Ziprasidone augmentation for anxious depression. Int Clin Psychopharmacol. 2016 Nov;31(6):341-6. doi: 10.1097/YIC.0000000000000133. PMID 27306192
- [Derived] Papakostas GI, Fava M, Baer L, Swee MB, Jaeger A, Bobo WV, Shelton RC. Ziprasidone Augmentation of Escitalopram for Major Depressive Disorder: Efficacy Results From a Randomized, Double-Blind, Placebo-Controlled Study. Am J Psychiatry. 2015 Dec;172(12):1251-8. doi: 10.1176/appi.ajp.2015.14101251. Epub 2015 Jun 18. PMID 26085041

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 458 patients met eligibility criteria for the study and were enrolled in an 8-week, open-label, flexible dose trial of escitalopram. At the end of this open-label trial, 139 patients not responding to Escitalopram were randomized to receive adjunctive ziprasidone or adjunctive placebo.
Groups:
- Ziprasidone + Escitalopram: Patients in group 1 will receive Ziprasidone added to Escitalopram for the full 8 weeks of Phase 2.
  Ziprasidone: 20mg-80mg a day. Dose increases of 20mg per day may occur at three study visits as directed by clinician. Maximum; 80mg per day per patient.
- Placebo + Escitalopram: Patients in group 2 will receive Placebo added to Escitalopram for the full 8 weeks of Phase 2.
  Placebo: 0mg Placebo per day (1-4 tablets per day). "Dose increases" and "dose decreases" may occur, but patient will remain at 0mg placebo.
Period: Overall Study
Arm/Group | Ziprasidone + Escitalopram | Placebo + Escitalopram
Started | 71 | 68
Completed | 49 | 53
Not Completed | 22 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziprasidone + Escitalopram | Placebo + Escitalopram | Total
Number analyzed (Participants) | 71 | 68 | 139
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.7 (13.8) | 44.2 (11.0) | 44.5 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 49 | 98
  Male | 22 | 19 | 41
Region of Enrollment [Number; unit: participants]
  United States | 71 | 68 | 139

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Will be Response Rates (50% Decrease in HAM-D-17 Scores) During Phase 2
Description: The primary outcome measure will be response rates (50% decrease in HAM-D-17 scores) during phase 2. A responder will be a patient who experiences a 50% or greater decrease in symptoms according to the HAM-D-17 during phase 2.
Time Frame: 8 Weeks
Measure: Number; unit: Percentage of patients
Arm/Group | Ziprasidone + Escitalopram | Placebo + Escitalopram
Number analyzed (Participants) | 71 | 68
Percentage of patients | 35.2 | 20.5

2. Secondary Outcome: Remission Rates (HAM-D 17 Scores of Less Than 8) After Treatment Phase 2.
Description: A secondary outcome measure will be remission rates (HAM-D 17 scores of less than 8) after treatment phase 2.. A remitted will be a patient with a final score of 7 or less on the HAMD-17 during phase 2.
Time Frame: 8 weeks
Measure: Number; unit: Percentage of patients
Arm/Group | Ziprasidone + Escitalopram | Placebo + Escitalopram
Number analyzed (Participants) | 71 | 68
Percentage of patients | 38 | 30

3. Secondary Outcome: Comparing Scores on HAM-D 17 Baseline Visit to Phase 2 Final Visit at Week 8
Description: This will involve looking at the change in HAM-D 17 scores during phase 2. For HAMD-17 the minimum is 0, the maximum is 52, and greater scores represent more symptoms.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone + Escitalopram | Placebo + Escitalopram
Number analyzed (Participants) | 71 | 68
units on a scale | -6.4 (6.4) | -3.3 (6.2)

ADVERSE EVENTS:
Groups:
- Ziprasidone + Escitalpram: Patients in group 1 will receive Ziprasidone for the full 8 weeks of Phase 2.
  Ziprasidone: 20mg-80mg a day. Dose increases of 20mg per day may occur at three study visits as directed by clinician. Maximum; 80mg per day per patient.
- Ziprasidone + Placebo: Patients in group 2 will receive Placebo for the full 8 weeks of Phase 2.
  Placebo: 0mg Placebo per day (1-4 tablets per day). "Dose increases" and "dose decreases" may occur, but patient will remain at 0mg placebo.
Arm/Group | Ziprasidone + Escitalpram | Ziprasidone + Placebo
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/68
Other Adverse Events (participants affected / at risk) | 51/71 | 42/68
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ziprasidone + Escitalpram (N=71) | Ziprasidone + Placebo (N=68)
Somnolence and/or Fatigue (Nervous system disorders) | 24 (24) | 8 (8)
Akathisia (Nervous system disorders) | 11 (11) | 5 (5)
Headaches (Nervous system disorders) | 5 (5) | 9 (9)
Irritability (Nervous system disorders) | 7 (7) | 1 (1)
Poor concentration and/or memory (Nervous system disorders) | 6 (6) | 1 (1)
Insomnia (Nervous system disorders) | 6 (6) | 6 (6)
Dizziness (Nervous system disorders) | 5 (5) | 3 (3)
Anxiety and/or Agitation (Nervous system disorders) | 4 (4) | 0 (0)
Muscle Twitching (Nervous system disorders) | 8 (8) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 7 (7) | 11 (11)
Nausea (Gastrointestinal disorders) | 3 (3) | 9 (9)
GI Upset (Gastrointestinal disorders) | 8 (8) | 3 (3)
Sexual Dysfunction (Nervous system disorders) | 7 (7) | 5 (5)
Weight Gain (Metabolism and nutrition disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No